CLINICAL TRIAL: NCT00258180
Title: High-Dose Cyclophosphamide for the Treatment of Severe Autoimmune Enteropathy
Brief Title: Cyclophosphamide in Treating Young Patients With Severe Autoimmune Enteropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 03-07-08-04; P30CA006973 (NIH); JHOC-J0326 (Other: SKCCC); J0326 (Other: SKCCC); CDR0000441133 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Diarrhea; Gastrointestinal Complications; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; gastrointestinal complications; diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide

ARMS (1):
- severe autoimmune enteropathy (Experimental): Young patients with severe autoimmune enteropathy receive cyclophosphamide IV over 1 hour on days 1-4. Patients then receive filgrastim (G-CSF) IV or subcutaneously once daily beginning on day 10 and continuing for 3 days or until blood counts recover
  Interventions: Biological: filgrastim; Drug: cyclophosphamide

INTERVENTIONS:
Biological: filgrastim — Administered IV or subcutaneously once daily beginning on day 10 and continuing for 3 days or until blood counts recover
  Other Names: G-CSF
Drug: cyclophosphamide — Administered IV over 1 hour on days 1-4

SUMMARY:
RATIONALE: Cyclophosphamide may help control the symptoms of autoimmune enteropathy .

PURPOSE: This phase II trial is studying how well cyclophosphamide works in treating young patients with severe autoimmune enteropathy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of treatment-free remission in young patients with severe autoimmune enteropathy treated with high-dose cyclophosphamide.

Secondary

* Determine the toxic effects of this drug in these patients.

OUTLINE: Patients receive cyclophosphamide IV over 1 hour on days 1-4. Patients then receive filgrastim (G-CSF) IV or subcutaneously once daily beginning on day 10 and continuing for 3 days or until blood counts recover.

After completion of study treatment, patients are followed periodically for up to 1½ years.

PROJECTED ACCRUAL: A total of 7-11 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of severe autoimmune enteropathy

  * Condition is resistant to conventional therapy
* Histologic evidence of severe villous atrophy with intense lymphocytic infiltrate of the lamina propria by small intestinal biopsy within the past 3 months
* Disease failed to respond after ≥ 2 months of corticosteroid therapy at a dose of ≥ 0.5 mg/kg/day or ≥ 40 mg/day for patients > 20 kg AND 1 of the following therapies:

  * Cyclosporine resulting in ≥ 1 whole blood level of > 200 ng/mL
  * Tacrolimus resulting in ≥ 1 whole blood level of 5 ng/mL
* At least 50% estimated caloric needs provided by parenteral nutrition
* History of intractable diarrhea, defined as frequent watery stools for > 3 months that does not respond to dietary restriction
* No celiac disease, defined by a history of positive antiendomysial antibody or tissue transglutaminase antibody
* No primary immunodeficiency or x-linked autoimmunity-allergy dysregulation

PATIENT CHARACTERISTICS:

Performance status

* Lansky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* Ejection fraction ≥ 40% OR shortening fraction ≥ 20%

Pulmonary

* FVC or FEV_1 ≥ 50% of predicted (for patients > 8 years of age)
* No clinically abnormal pulmonary function or abnormal pulse oximetry (for patients ≤ 8 years of age)

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 9 months after completion of study treatment
* No known chromosomal abnormality

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No immunizations for at least 6 months after completion of study treatment

Endocrine therapy

* See Disease Characteristics
* At least 5 days since prior corticosteroids
* No concurrent dexamethasone as an anti-emetic

Other

* At least 5 days since other prior immunosuppressive medications (e.g., tacrolimus or cyclosporine)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2005-08-15 (Actual); Primary Completion 2009-02-24 (Actual); Study Completion 2009-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Loeb, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Maria Oliva-Hemker, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject was not assigned intervention due to PI decision.
Period: Overall Study
Arm/Group | Severe Autoimmune Enteropathy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Severe Autoimmune Enteropathy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-free Remission at 1 Year After Study Completion
Description: Number of participants off therapy 1 year after study completion without relapse.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Autoimmune Enteropathy
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: Number of Participants Experiencing Intervention-related Adverse Events, as Defined by CTCAE at 1 Month
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Autoimmune Enteropathy
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 1 year post-intervention
Arm/Group | Severe Autoimmune Enteropathy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No